CLINICAL TRIAL: NCT00431951
Title: Double-blind, Randomized, Placebo-controlled, Escalating, Multiple-dose, Phase I Trial to Assess Safety, Tolerability and Pharmacokinetics of ST-246 Administered as a Single Daily Dose for 21 Days in Healthy, Non-fasted Volunteers
Brief Title: Phase I, Escalating, Multiple-Dose, ST-246 Safety, Tolerability and Pharmacokinetics 21-Day Trial in Healthy Volunteers
Acronym: SIGA-246-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SIGA Technologies (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ST-246 RD PHS 1; DMID 06-0080 (Other: NIH Contract #: HHSN266200600014C)
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Results first posted 2010-05-07 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — tecovirimat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ST-246 (Experimental): 250 mg, 400 mg or 800 mg of ST-246 given once daily for 21 days
  Interventions: Drug: ST-246
- placebo (Placebo Comparator): Placebo to match ST-246
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ST-246 — 250 mg, 400 mg or 800 mg capsules given once daily for 21 days
  Other Names: Tecovirimat
  Arms: ST-246
Drug: Placebo — Capsules to match experimental drug
  Other Names: Placebo to match ST-246
  Arms: placebo

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and pharmacokinetics of a single, daily, oral dose of ST-246 (either 250, 400 or 800mg) administered for 21 days to 30 healthy, fed volunteers.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled, dose-escalating, multiple-dose study of orally administered ST-246 to 30 healthy volunteers ages 18-50 years, randomized to receive either active drug (8 subjects) or placebo (2 subjects) in 1 of 3 dosing groups (250, 400 or 800mg groups). Each dose group of 10 was divided into two cohorts of 5 subjects (4 active and 1 placebo). The first cohort was dosed approximately 4-8 weeks before the second cohort of each dose group. Dose groups completed the study treatment approximately 5 weeks prior to the start of the following dose group. Study procedures included several overnight stays, medical history/exam, laboratory testing done by blood draw, and electrocardiograms.

ELIGIBILITY:
Subject Inclusion Criteria:

* Healthy volunteers
* Ability to Consent
* Not taking any other medication
* Adequate venous access
* Using adequate birth control

Subject Exclusion Criteria:

* Inability to swallow study medication.
* Pregnant or breastfeeding
* Received experimental drug within 30 days of study entry or will participate in any experimental study during the study period.
* Current drug abuse, alcohol abuse, or homelessness.
* Taking concomitant medication
* Lactose Intolerance
* Medical condition; e.g., asthma, diabetes, thyroid disease, angioedema, BMI >35 or <18, hypertension, bleeding disorder, malignancy, seizure, neutropenia, Hepatitis B or C, HIV or AIDS.
* Any condition, occupational reason or other responsibility that, in the judgment of the Investigator, would jeopardize the safety or rights of a volunteer, or render the subject unable to comply with the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research
Locations (1):
- Orlando Clinical Research, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one site, Orlando Clinical Research Center, Orlando, FL. The study was conducted in healthy volunteers from the site's database.
Pre-assignment Details: After a 28-day screening and 1-day enrollment period, study drug was administered on Day 1. Ten participants (8 drug:2 placebo) were randomized in each of three dosing groups (250, 400, and 800 mg ST-246). Each group was divided into 2 cohorts of 5 subjects (4 drug:1 placebo), with one cohort receiving drug 4-8 weeks before the other cohort.
Groups:
- ST-246 250 mg: 250 mg ST-246 given as a single daily oral dose to 8 subjects for 21 days.
- ST-246 400mg: 400 mg ST-246 given as a single daily oral dose to 8 subjects for 21 days. Blood and urine samples for PK taken on Days 1, 6, and 21.
- ST-246 800 mg: 800 mg ST-246 given as a single daily oral dose to 8 subjects for 21 days. Blood and urine samples for PK taken on Days 1, 6, and 21.
- Placebo: Placebo given as a single daily oral dose for 21 days to 6 subjects, to match ST-246 doses (2 patients for each dose equivalent). Blood and urine samples for PK taken on Days 1, 6, and 21.
Period: Overall Study
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Started | 8 | 8 | 8 | 6
Completed | 7 | 6 | 6 | 4
Not Completed | 1 | 2 | 2 | 2
Not completed — Inability to follow study procedures | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 6 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.2) | 27.6 (7.8) | 37.5 (7.6) | 34.8 (8.9) | 33.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 2 | 10
  Male | 5 | 4 | 7 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Who Tolerated ST-246 (250, 400 or 800mg) as Determined by Changes in Safety Parameters, According to the Division of Acquired Immunodeficiency Syndrome (DAIDS) Adverse Events (AE) Grading Table
Description: Evaluated safety parameters included:
  1. physical examination/vital signs
  2. electrocardiograms (heart rate, PR interval, QRS duration, QT interval, and QTc Bazett)
  3. laboratory safety tests (hematology, chemistry, urinalysis)
  4. adverse events (AEs) For a)-c), statistical values (mean, standard deviation, median, minimum, maximum) and changes from baseline (Day 1 pre-dose) to each time-point, were compared to laboratory normal reference ranges. If values for a)-d) were a Grade 3 or higher (in DAIDS AE Table)and ST-246-related, they were considered severe and significant, respectively.
Time Frame: Days 1, 6, 14-16, 21-24, 28-31, and 51-53
Population: Post-screening, 30 healthy subjects were randomized into three active drug groups with 8 subjects each, and one placebo group with 6 subjects. A total of 7 withdrawals during the entire study were due to inability to follow procedure (4), lost to follow-up (1), requested due to concomitant medication (1), and an adverse event (1)
Measure: Number; unit: Participants
Groups:
- ST-246 400mg: 400 mg ST-246 given as a single daily oral dose to 8 subjects for 21 days.
- ST-246 800 mg: 800 mg ST-246 given as a single daily oral dose to 8 subjects for 21 days.
- Placebo: Placebo given as a single daily oral dose for 21 days to 6 subjects, to match ST-246 doses (2 patients for each dose equivalent).
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
Participants | 8 | 8 | 7 | 6

2. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Cmax
Description: Cmax: Maximum drug concentration in plasma determined directly from individual concentration-time data
Time Frame: Day 1
Population: Post-screening, 30 healthy subjects were randomized on Day 1 into three active drug groups with 8 subjects each and one placebo group with 6 subjects
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ST-246 250 mg: 250 mg ST-246 given as a single daily oral dose to 8 subjects for 21 days. Blood and urine samples for PK taken on Days 1, 6, and 21.
- Placebo: Placebo given as a single daily oral dose to 6 subjects for 21 days, to match ST-246 doses (2 patients for each dose equivalent). Blood and urine samples for PK taken on Days 1, 6, and 21.
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
ng/mL | 985 (346) | 1392 (411) | 2279 (395) | 0 (0)

3. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Cmax
Description: Cmax: Maximum drug concentration in plasma determined directly from individual concentration-time data
Time Frame: Day 6
Population: Post-screening, 30 healthy subjects were randomized into three active drug groups with 8 subjects each and one placebo group with 6 subjects. By Day 6 there were 3 (out of 7 total) withdrawals from the study due to inability to follow procedure (2; 800mg and placebo groups), and requested due to concomitant medication (1; 400mg group)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 7 | 5
ng/mL | 1212 (350) | 1298 (277) | 2337 (437) | 0 (0)

4. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Cmax
Description: Cmax: Maximum drug concentration in plasma determined directly from individual concentration-time data
Time Frame: Day 21
Population: Post-screening, 30 healthy subjects were randomized into three active drug groups with 8 subjects each and one placebo group with 6 subjects. Between Days 6 and 21, there were 4 (out of 7 total) withdrawals due to inability to follow procedure (2; 250mg and placebo groups), lost to follow-up (1; 400mg group), and adverse event (1; 800mg group)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 4
ng/mL | 1101 (378) | 1457 (451) | 2437 (496) | 0 (0)

5. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Tmax
Description: Tmax: Time to reach maximum drug concentration in plasma calculated from [plasma] versus time profiles.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
hours | 3.0 (1.1) | 3.3 (1.0) | 2.9 (1.3) | 0 (0)

6. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Tmax
Description: Tmax: Time to reach maximum drug concentration in plasma calculated from [plasma] versus time profiles.
Time Frame: Day 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 7 | 5
hours | 2.6 (1.2) | 3.7 (2.1) | 3.6 (2.3) | 0 (0)

7. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Tmax
Description: Tmax: Time to reach maximum drug concentration in plasma calculated from [plasma] versus time profiles.
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 4
hours | 2.9 (1.1) | 2.7 (1.0) | 3.2 (1.3) | 0 (0)

8. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: t½
Description: t½: Observed terminal elimination half-life determined after the last dose on Day 21
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 4
hours | 18.8 (10.4) | 19.9 (8.9) | 20.7 (8.4) | 0 (0)

9. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: AUCtau
Description: AUCtau: Area under the plasma concentration-time curve for each dosing interval (from time 0 to 24 hours sample) determined using the linear trapezoidal rule
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
ng*hr/mL | 9101 (3492) | 13146 (3626) | 20959 (6091) | 0 (0)

10. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: AUCtau
Description: as for outcome 9
Time Frame: Day 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 7 | 5
ng*hr/mL | 11892 (4389) | 15432 (4708) | 23352 (4696) | 0 (0)

11. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: AUCtau
Description: as for outcome 9
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 4
ng*hr/mL | 10083 (2843) | 16182 (5534) | 22684 (4579) | 0 (0)

12. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Ae(0-24)
Description: Ae(0-24): Cumulative amount of drug excreted unchanged in urine over 24 hours (three 8-hour collection periods), determined on Days 1 and 21
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
mg | 0.041 (0.031) | 0.110 (0.066) | 0.157 (0.048) | 0 (0)

13. Secondary Outcome: Evaluation of Pharmacokinetic Parameters to Assess Interventions: Ae(0-24)
Description: as for outcome 12
Time Frame: Day 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 4
mg | 0.049 (0.026) | 0.108 (0.046) | 0.213 (0.165) | 0 (0)

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: Study drug was administered to each dosing group cohort for 21 days and subjects were followed for an additional 30 to 32 days. AEs were recorded throughout this time period.
Arm/Group | ST-246 250 mg | ST-246 400mg | ST-246 800 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 6/8 | 2/8 | 5/8 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST-246 250 mg (N=8) | ST-246 400mg (N=8) | ST-246 800 mg (N=8) | Placebo (N=6)
Abnormal Eye Sensation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Backpain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 4 (4) | 2 (2) — Only one subject, in the 800mg group, experienced a severe headache (TEAE of Grade 3; deemed study-drug related) on Day 15, and discontinued the study.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must obtain the sponsor's written consent to publish any study results and must notify the sponsor within 30 working days prior to publishing.